CLINICAL TRIAL: NCT04240977
Title: Feasibility and Single-arm Trial of HOBSCOTCH Telehealth Intervention in Refractory Epilepsy
Brief Title: Feasibility of HOBSCOTCH Telehealth Intervention in Refractory Epilepsy
Acronym: HOBSCOTCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: L -1063-19; 90SFGE0010 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2019-12-17; First posted 2020-01-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Refractory Epilepsy
Keywords: Refractory epilepsy, self-management; Quality of life
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: This study utilizes a single-arm pre/post experimental design with an additional 3-month maintenance assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Behavioral: HOBSCOTCH: "Home-Based Self-Management and Cognitive Training Changes Lives"

INTERVENTIONS:
Behavioral: HOBSCOTCH: "Home-Based Self-Management and Cognitive Training Changes Lives" — Home-Based Self-Management and Cognitive Training Changes Lives (HOBSCOTCH) is a novel phone-based intervention that is enables acquisition of cognitive skills in line with problem solving therapy (PST), and is well suited for PWRE who have failed all other treatment alternatives. Sessions #2 through #7 focus on building patient's awareness for their own day-to-day memory problems, brainstorming, implementing and reviewing the outcomes of potential solutions they generate themselves using the PST framework. In each of these sessions, providers will assist patients in generating alternative solutions, in thinking through what the implementation of each strategy would entail, and in helping them review outcomes for adopted strategies to refine their approach for optimized adoption and generalization.

SUMMARY:
The purpose of this study is to see whether a phone-intervention called HOBSCOTCH will improve health, daily functioning and quality of life among patients with refractory epilepsy. HOBSCOTCH stands for "Home-Based Self-Management and Cognitive Training Changes Lives." This study will also help to find the best ways of integrating this telehealth intervention to routine clinic use.

DETAILED DESCRIPTION:
The proposed project will assess the efficacy of an 8-week phone-delivered, experimental treatment called "Home-Based Self-Management and Cognitive Training Changes Lives" (HOBSCOTCH) on sixty patients with refractory epilepsy (PWRE). The investigators will employ a prospective, single blind randomized clinical trial design with wait-list controls to examine both objective and subjective measures of daily life, daily functioning, cognition, and emotional well-being. Investigators will also assess the impact of HOBSCOTCH on employment and work productivity using the Lam Employment absence and Disability Scale (LEAPS) and the Sheehan Disability Scale (SDS). Lastly, the investigators will examine whether changes in these domains are maintained three months after completion of the intervention. The study will expand the efficacy literature for HOBSCOTCH and further refine its use in a busy clinical environment, and therefore has potential to benefit the patient population (PWRE), who currently lacks treatment options besides the pharmacological and surgical care currently available.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read and speak English.
* Patient has a reliable telephone connection and a private place they can use during the course of this study
* They do not have any treatment or intervention plan in place for the next 6 months. They may be on an anti-epileptic drug regimen that has not been changed in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life in Epilepsy - 31 score | baseline & 8-10 weeks after baseline
  overall raw score [15-97] that corresponds to reported levels of worry, emotional well-being, energy/fatigue, cognitive functioning, medication effects and social functioning

SECONDARY OUTCOMES:
Feasibility of HOBSCOTCH in the clinical setting | baseline
  Physicians involved (count), referrals made (count), patients contacted and screened (count), patients enrolled (count), patient completing the intervention (count)

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No individual level data will be shared.